CLINICAL TRIAL: NCT04718090
Title: Comparison of Postoperative Analgesic Consumption and Pain in Shoulder Surgery Patients Undergoing Interscalene and Pericapsular Nerve Group (PENG) Blocks
Brief Title: Comparison of Interscalene and Pericapsular Nerve Group (PENG) Block in Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Collaborators: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Merve Yazici Kara, M.D., Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MYaziciKara-1
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Visual Analogue Score

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interscalene block (Active Comparator)
  Interventions: Procedure: PENG Block
- PENG block (Active Comparator)
  Interventions: Procedure: PENG Block

INTERVENTIONS:
Procedure: PENG Block — Pericapsular nerve group block in shoulder surgery.

SUMMARY:
Early postoperative pain after shoulder surgery is a major concern and distress for patients and orthopedic surgeons. Adequate pain control; It is vital for all aspects of patient recovery, including mental state, nutrition, cost of care period, rehabilitation, patient satisfaction, and overall post-surgery outcomes.Single analgesic regimens are not always effective in controlling moderate to severe postoperative pain.Therefore, multimodal pain management is preferred and is currently recommended for early postoperative pain control.Regional anesthesia is preferred in shoulder surgery as an effective way to provide anesthesia and postoperative analgesia.To ensure adequate postoperative pain control, nerve supply to the synovium, capsule, joint surfaces, ligaments, periosteum and shoulder muscles must be blocked.Interscalene blocks are well studied and established means of providing analgesia following shoulder surgery and are considered the gold standard mode of regional anesthesia.Pericapsular nerve group block is a new block that provides a pericapsular distribution with local anesthetic infiltration around the glenohumeral joint and provides analgesia without motor blockage by reaching the sensory nerve branches of the glenohumeral joint.The aim of this study was to compare the results between interscalene block and pericapsular nerve group block in patients undergoing shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* American Society of Anesthesiologists (ASA) 1 and 2
* shoulder surgery

Exclusion Criteria:

* under 18 years old
* American Society of Anesthesiologists (ASA) 3 and above
* who are allergic to local anesthetics
* patients with infection at the injection site
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 5 months
  Visual Analogue Scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Patel MS, Abboud JA, Sethi PM. Perioperative pain management for shoulder surgery: evolving techniques. J Shoulder Elbow Surg. 2020 Nov;29(11):e416-e433. doi: 10.1016/j.jse.2020.04.049. Epub 2020 Jun 9. PMID 32844751
- [Result] Sripada R, Bowens C Jr. Regional anesthesia procedures for shoulder and upper arm surgery upper extremity update--2005 to present. Int Anesthesiol Clin. 2012 Winter;50(1):26-46. doi: 10.1097/AIA.0b013e31821a0284. PMID 22227421
- [Result] Yamak Altinpulluk E, Teles AS, Galluccio F, Simon DG, Olea MS, Salazar C, Fajardo Perez M. Pericapsular nerve group block for postoperative shoulder pain: A cadaveric radiological evaluation. J Clin Anesth. 2020 Dec;67:110058. doi: 10.1016/j.jclinane.2020.110058. Epub 2020 Sep 26. No abstract available. PMID 32987232
- [Result] Tran J, Peng PWH, Agur AMR. Anatomical study of the innervation of glenohumeral and acromioclavicular joint capsules: implications for image-guided intervention. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100152. doi: 10.1136/rapm-2018-100152. Online ahead of print. PMID 30635516